CLINICAL TRIAL: NCT05365633
Title: Empowering Sexual and/or Gender Minority Tobacco Cessation: A Pilot Study
Brief Title: Empowering LGBTQ+ Tobacco Cessation Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14472
Record Dates: First submitted 2022-04-12; First posted 2022-05-09 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
Keywords: sexual and gender minorities; LGBT; empowerment; tobacco use; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Coitus; Empowerment; Tobacco Use

STUDY DESIGN:
Intervention Model Description: Single-arm pilot design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empowerment activity-enhanced tobacco cessation assistance (Other): Single arm pilot intervention design to assess feasibility and acceptability
  Interventions: Behavioral: Empowerment activity-enhanced tobacco cessation assistance

INTERVENTIONS:
Behavioral: Empowerment activity-enhanced tobacco cessation assistance — Participants will receive standard Tobacco Treatment Research Program (TTRP) tobacco cessation assistance either remotely or in-person: 6 weekly counseling sessions and 12 weeks of combination NRT (nicotine patches + nicotine gum or lozenges). During the 6 weeks of counseling, participants will also engage in at least 4 'empowerment activities' (i.e., SGM social change mobilization and community-building activities48) for a total of at least 8 hours. Activities will be tailored to each participant's comfort level and skills. Examples are compiling publicly-available information about school board meetings to support community members in participating in their school districts and making follow-up phone calls with a script to Freedom OK's name change clinic participants.

SUMMARY:
Sexual and/or gender minority (SGM) people have disproportionately high rates of tobacco use - the number one cause of preventable death. Reasons for this include using tobacco to cope with social minority stressors, pro-tobacco use norms in SGM social spaces and networks, and targeted tobacco industry marketing. Empowerment Theory explains how positive behavior change, like quitting smoking, can be promoted through skills development with greater participation in the public affairs of one's community. An empowerment approach may enhance tobacco cessation treatment for SGM people and other stigmatized groups because it links individual well-being with the larger social and political context. This pilot study will assess the acceptability, feasibility, and preliminary impact of empowerment-enhanced tobacco smoking cessation assistance for SGM adults. We will enroll N=20 SGM adults in Oklahoma who smoke and are willing to quit. Participants will receive standard tobacco cessation assistance through the Stephenson Cancer Center Tobacco Treatment Research Program (TTRP). Concurrently, they will also engage in 'empowerment activities', meaning SGM organizing and community-building activities, like conducting follow-up phone calls to name change clinic participants. This will be guided by an Oklahoman SGM-serving community partner. Participants will complete 8 surveys during the intervention period and 12 weeks post-quit-date, a 60-minute, in-depth exit interview, and biochemically-verified smoking status before the intervention and 12 weeks post-quit-date. This pilot study will establish collaborative relationships between the PI's team and local SGM-serving organizations, and will produce preliminary findings to support future R01-level funding to conduct a fully-powered randomized control trial of a multi-level empowerment-enhanced SGM tobacco cessation intervention.

DETAILED DESCRIPTION:
Aim 1: Assess the feasibility and acceptability of empowerment-enhanced tobacco cessation assistance for sexual and/or gender minority (SGM) adults. Use baseline and exit surveys and in-depth interviews to assess retention, empowerment activity participation (e.g., number, duration, intensity, roles), and participants' perceptions of the intervention.

Aim 2: Compare individual empowerment and cessation predictors pre- and post-intervention. Hypothesis: Post intervention, participants will have (i) increased adaptive coping strategies, social support, and smoking abstinence self-efficacy; and (ii) decreased internalized SGM stigma.

Aim 3: Assess tobacco cessation outcomes post-intervention. Hypothesis: The proportion of participants with biochemically-verified smoking abstinence at 12 weeks post-quit-date will be equal to or greater than the general Stephenson Cancer Center Tobacco Treatment research Program (TTRP) intervention (i.e., 18% biochemically-verified abstinence at 12 weeks1); medication and counseling adherence will be moderate/optimal for >50% of treatment weeks.

Study overview. This study will assess the feasibility and acceptability of empowerment-enhanced tobacco cessation assistance for SGM adults. A single-arm pilot design will be used given funding, time, and sampling pool limits. Participants (N=20) will receive standard TTRP tobacco cessation assistance and concurrently participate in SGM empowerment activities. Outcomes will be assessed quantitatively and qualitatively. Primary outcome variables will be retention, perceptions of the intervention, adaptive coping strategies, biochemically-verified smoking abstinence at 12 weeks post-quit-date, and treatment adherence.

Recruitment. Participants will be enrolled over a 4-month period and recruit through the TTRP, which serves an average of 30 SGM individuals per year without SGM-targeted recruitment. This will be supplement by recruiting via local SGM-serving organizations, SGM targeted social media ads (e.g., Facebook), and snowball recruitment.

Intervention. Participants will receive standard TTRP tobacco cessation assistance either remotely or in-person: 6 weekly counseling sessions and 12 weeks of combination NRT (nicotine patches + nicotine gum or lozenges). During the 6 weeks of counseling, participants will also engage in at least 4 'empowerment activities' (i.e., SGM social change mobilization and community-building activities48) for a total of at least 8 hours. Activities will be tailored to each participant's comfort level and skills. Examples are compiling publicly-available school board information to make it easier for community members to participate in their school districts and follow-up phone calls to Freedom OK's name correction clinic participants.

Participants will complete the following assessments: (i) 8 surveys (baseline, exit, quit-day, 1-4 and 12 weeks post-quit-date); (ii) biochemically-verified smoking status at baseline and 12 weeks post-quit-date via expired carbon monoxide monitors; and (iii) a 60-minute in-depth interview over Zoom video chat within weeks 6-8 post-quit-date. Participants will be incentivized a total of $200 for the baseline survey ($25), 6 subsequent surveys ($70), 2 expired carbon monoxide tests ($20), exit survey ($25), and 60-minute interview ($60). Freedom Oklahoma staff will participate in interviews and reflect on the intervention and Freedom OK's role in it. Freedom Oklahoma will adopt a tobacco-free policy and provide feedback on the cultural competence of TTRP materials.

Partnerships. TTRP will provide the standard tobacco cessation assistance. Freedom Oklahoma will design the empowerment activities. Freedom Oklahoma is a community-based organization in Oklahoma City that has worked to secure lived equality and legal protection for SGM Oklahomans for over 15 years. PI McQuoid and Freedom OK have held more than 4 project planning meetings over the past year.

Measurement of Feasibility and Acceptability (Aim 1). Exit surveys administered via REDCap will be used to assess retention and self-reported empowerment activity participation (i.e., total hours, types of events/activities, roles played).73 This will be cross-referenced with research project records of empowerment activity participation. Perceptions of the intervention will be qualitatively assessed by interviewing participants over Zoom video chat at 12 weeks post-quit-date. PI McQuoid, a qualitative methods expert, will train a team to conduct semi-structured, in-depth interviews lasting approximately 60 minutes. Rich content will be elicited regarding experiences of empowerment activity participation and tobacco cessation as an SGM person in Oklahoma. Interview guide domains will include: (i) best intervention aspects (e.g. highlights, peak experiences); (ii) biggest challenges or negative experiences; (iii) empowerment activity experiences; (iv) interactions of empowerment activity participation with tobacco cessation experiences; (v) outcomes and personal growth (vi) suggestions for intervention improvements. Interviews will be audio-recorded and professionally transcribed verbatim.

Qualitative Analysis: Dedoose qualitative data analysis software will be used to conduct an inductive-deductive thematic transcript analysis with a priori themes derived from ET and SGM tobacco cessation literature.33-35 An iterative codebook development process will be used involving weekly team discussions, independent coding, and member checking of findings74 to enhance rigor and trustworthiness.75,76 Freedom Oklahoma staff will also be interviewed about their perceptions of the intervention and their organization's role in it.

Measurement of Individual Empowerment and Cessation Predictors (Aim 2). Individual empowerment and cessation predictors pre- and post-intervention will be compared with baseline and exit surveys. Predictors of smoking cessation51-54,77,78 and individual empowerment outcome measures will be compared, adapted from a youth empowerment tobacco control model42,73 and SGM social change mobilization participation research.48 These will include: (i) adaptive coping strategies (Cognitive Emotion Regulation Questionnaire79), (ii) (v) social support (Relational Health Indices80), (iii) abstinence self-efficacy (Confidence Inventory81), and (iv) internalized SGM stigma (Internalized Transphobia and Pride82 and Internalized Homophobia items83).

Measurement of Tobacco Cessation Outcomes (Aim 3). Benchmarks will be used to assess participants' tobacco cessation outcomes. Tobacco abstinence will be measured via self-report and biochemically-verified via expired carbon monoxide at baseline and 12 weeks post-quit-date. Treatment adherence will be assessed with the 4-item Medication Adherence Questionnaire (MAQ)84 and counseling session attendance tracking.

Sample Size/Analysis Plan. Primary outcome variables will be: retention, perceptions of the intervention, adaptive coping strategies, biochemical verification of tobacco abstinence at 12 weeks post-quit-date, and treatment adherence. Retention will be evaluated by calculating the proportion of participants who complete the final study visit at 12-weeks post-quit, with the goal of retaining >80% of participants. Perceptions of the intervention will be qualitatively evaluated (as described above). A two-sided paired samples t-test will be used to examine the mean differences in adaptive coping strategies pre- and post-intervention (α=0.05). Assuming 20% attrition and a standard deviation of differences of 4.085, n=20 participants will provide 80% power to detect a mean difference of 2.6 in adaptive coping strategies. Tobacco cessation outcomes will be considered successful if the proportion of participants with biochemically-verified smoking abstinence (expired carbon monoxide) at 12 weeks post-quite-date is equal to or greater than the general TTRP sample (i.e., 18% at 12 weeks1). Treatment adherence will be considered successful with all participants having >50% of treatment weeks with an MAQ score indicating moderate/high adherence and counseling session attendance.

Expected outcomes: Empowerment-enhanced tobacco cessation assistance will be acceptable and feasible (Aim 1), will increase within-subject empowerment and improve cessation predictors (Aim 2), and will meet benchmarks for tobacco cessation outcomes (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Self-identify as sexual and/or gender minority
* Reside in the State of Oklahoma
* Report past 30 day use of combustible tobacco
* Willing to quit using combustible tobacco within the next 2 weeks
* English-speaking
* Willing to refrain from smoking any substance, such as cannabis, within 48 hours of expired carbon monoxide collection
* Willing to complete all intervention components and data collection activities

Exclusion Criteria:

* Have contraindications for nicotine replacement therapy (NRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia McQuoid, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available to outside investigators upon request. However, it is noteworthy that data collected as part of the current proposal will be from a small sample, and will not provide sufficient information from which to draw conclusions. Rather these data will support a larger, adequately powered trial, from which data may be more complete and useful to other investigators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited online from Oklahoma and consented online August 2022 - September 2023.
Pre-assignment Details: 20 participants signed consent, were fully enrolled, and were randomized to the intervention.
Period: Overall Study
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Started | 20 (20 individuals started the intervention (i.e., they completed at least one smoking cessation counseling session or volunteering session); these 20 comprise the analytic sample.)
Completed | 16 (16 completed the intervention, meaning they completed an exit survey at the end of the 12 week intervention period.)
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Empowerment Activity-enhanced Tobacco Cessation Assistance: Single arm pilot intervention design to assess feasibility and acceptability
  Empowerment activity-enhanced tobacco cessation assistance: Participants will receive standard Tobacco Treatment Research Program (TTRP) tobacco cessation assistance either remotely or in-person: 6 weekly counseling sessions and 12 weeks of combination nicotine replacement therapy (NRT); nicotine patches + nicotine gum or lozenges). During the 6 weeks of counseling, participants will also engage in at least 4 'empowerment activities' (i.e., SGM social change mobilization and community-building volunteer activities) for a total of at least 8 hours. Activities will be tailored to each participant's comfort level and skills. Examples are compiling publicly-available information about school board meetings to support community members in participating in their school districts and making follow-up phone calls with a script to Freedom OK's name change clinic participants.
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39.5 [30.0 to 47.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 4
    Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 15
  Race: Black/African American | 1
  Race: Indigenous Peoples, Native American, Alaskan Native | 3
  Race: Middle Eastern or North African | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: We will evaluate retention by calculating the proportion of participants who complete the final study visit at 12-weeks post-quit, with the goal of retaining >80% of participants.
Time Frame: 12-weeks post-quit
Population: Treatment group in a single-arm pilot trial
Measure: Count of Participants; unit: Participants
Groups:
- Empowerment Activity-enhanced Tobacco Cessation Assistance: Single arm pilot intervention design to assess feasibility and acceptability
  Empowerment activity-enhanced tobacco cessation assistance: Participants will receive standard Tobacco Treatment Research Program (TTRP) tobacco cessation assistance either remotely or in-person: 6 weekly counseling sessions and 12 weeks of combination NRT (nicotine patches + nicotine gum or lozenges). During the 6 weeks of counseling, participants will also engage in at least 4 'empowerment activities' (i.e., SGM social change mobilization and community-building activities48) for a total of at least 8 hours. Activities will be tailored to each participant's comfort level and skills. Examples are compiling publicly-available information about school board meetings to support community members in participating in their school districts and making follow-up phone calls with a script to Freedom OK's name change clinic participants. follow-up surveying of Freedom OK's name and gender marker change clinic72 participants.
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 20
Participants | 16

2. Primary Outcome: Number of Participants Endorsing That They Would Recommend This Intervention to Another LGBTQ2S+ Identified Person Who Wants to Quit Smoking
Description: Intervention acceptability will be assessed by the participant endorsing that they would recommend this intervention to another LGBTQ2S+ identified person who wants to quit smoking.
Time Frame: 12 weeks post-quit-date
Population: Participants who completed an exit survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 16
Participants | 13

3. Primary Outcome: Number of Community Partner Staff Who Perceived Their Organization's Partnership on the Intervention as Beneficial
Description: We will qualitatively assess community partner perceptions of their organization's partnership on the intervention as beneficial by interviewing Freedom Oklahoma staff over Zoom video chat. Semi-structured, in-depth interview lasting approximately 60 minutes will discuss Freedom Oklahoma staff's perceptions of the intervention and their organization's role in it.
Time Frame: within 1 month of data collection completion
Population: Interviews were conducted with 2 staff members from the community partner organization.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 2
Participants | 2

4. Primary Outcome: Number of Participants Having Had ≥ 2 Weeks With Moderate to High Adherence to the Nicotine Patch Assessed With the 4-item Medication Adherence Questionnaire (MAQ)
Description: Treatment adherence will be assessed with the 4-item Medication Adherence Questionnaire (MAQ) and counseling session attendance tracking. The benchmark for satisfactory medication treatment adherence is having had ≥ 2 weeks with moderate to high adherence to the nicotine patch.
Time Frame: 12 weeks post-quit-date
Population: Participants who completed an exit survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 16
Participants | 11

5. Primary Outcome: Number of Participants Attending at Least 4 Smoking Cessation Counseling Sessions
Description: Counseling attendance will be assessed by tracking the proportion of counseling sessions attended by each participant by 12 weeks post-quit-date. The benchmark for satisfactory attendance is attending at least 4 counseling sessions.
Time Frame: 12 weeks post-quit-date
Population: Participants who completed an exit survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 16
Participants | 14

6. Primary Outcome: Number of Participants Attending at Least 4 Volunteer Sessions
Description: Volunteer session attendance will be assessed by tracking the proportion of sessions attended by each participant by 12 weeks post-quit-date. The benchmark for satisfactory attendance is attending at least 4 sessions.
Time Frame: 12 weeks post-quit-date
Population: Participants who completed an exit survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 16
Participants | 10

7. Secondary Outcome: Number of Participants Self-reporting 7-day Point Prevalence Abstinence at Week 12
Description: Participant self-report of smoking abstinence within the past 7 days upon intervention exit. Participants who did not complete an exit survey are assumed to be smoking (i.e., not abstinent) at week 12.
Time Frame: 12 weeks post-quit-date
Population: Participants who started the intervention by completing at least one volunteer session or at least one counseling session.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 20
Participants | 9

8. Secondary Outcome: Number of Participants for Whom Self-reported Smoking Abstinence is Biochemically-verified
Description: We will use benchmarks to assess participants' tobacco cessation outcomes. Biochemically-verified smoking status will be measured via expired carbon monoxide at 12 weeks post-quit-date. Tobacco cessation outcomes will be considered successful if the proportion of participants with biochemically-verified smoking abstinence (expired carbon monoxide) at 12 weeks post-quite-date is equal to or greater than the general Tobacco Treatment Research Program (TTRP) sample (i.e., 18% at 12 weeks).
Time Frame: 12 weeks post-quit-date
Population: Technical problems hindered biochemical verification. The iCOTM Smokerlyzer carbon monoxide monitor smartphone app was incompatible with a newer Android operating system used by at least 7 participants. The team attempted to verify abstinence using in-person carbon monoxide devices (Vitalograph Model 2900 BreathCOTM), but due to participants' remote locations, readings were only obtained for 8/16 exit survey respondents. Of those 8, 5 participants self-reported smoking abstinence at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 5
Participants | 4

9. Secondary Outcome: Number of Participants Who Reported an Increase in Adaptive Coping From Baseline to Exit
Description: We will compare within subject adaptive coping strategies with baseline and exit surveys (12 weeks post-quit-date) using the Cognitive Emotion Regulation Questionnaire79. We will use a two-sided paired samples t-test to examine the mean differences in adaptive coping strategies pre- and post-intervention (α=0.05). Assuming a standard deviation of differences of 4.085, n=20 participants will provide 80% power to detect a mean difference of 2.6 in adaptive coping strategies.
Time Frame: baseline and 12 weeks post-quit-date
Population: Participants who completed an exit survey at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
Number analyzed (Participants) | 16
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov Definitions.
Groups:
- Empowerment Activity-enhanced Tobacco Cessation Assistance: Single arm pilot intervention design to assess feasibility and acceptability
  Empowerment activity-enhanced tobacco cessation assistance: Participants will receive standard Tobacco Treatment Research Program (TTRP) tobacco cessation assistance either remotely or in-person: 6 weekly counseling sessions and 12 weeks of combination NRT (nicotine patches + nicotine gum or lozenges). During the 6 weeks of counseling, participants will also engage in at least 4 'empowerment activities' (i.e., SGM social change mobilization and community-building activities48) for a total of at least 8 hours.
Arm/Group | Empowerment Activity-enhanced Tobacco Cessation Assistance
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT05365633/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT05365633/SAP_001.pdf